CLINICAL TRIAL: NCT05498493
Title: Assessing the Effectiveness of Cognitive Rehabilitation for Post-COVID-19 Cognitive Impairment: a Pilot Study
Brief Title: Cognitive Rehabilitation for Post-COVID-19 Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Juan Wisnivesky, Chief, Division of General Internal Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-20-00857
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Rehabilitation (Experimental): Active Group participants will receive nine 1.5-h sessions of virtual (via Zoom platform) group-based training, three individual virtual 1-h training sessions, and approximately 20 h of home practice and CCT over 12 weeks.
  Interventions: Behavioral: Cognitive Rehabilitation
- Brain Health Education Program (Active Comparator): The control group format will be twelve 1.5 or 1 h virtual sessions over 12 weeks, in addition to 20 h of home practice of a computerized control program (e.g., consisting of publicly available computer games such as sudoku and crossword puzzles).
  Interventions: Behavioral: Brain Health Education Program

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — The virtual small group format will include two to five participants and one facilitator per group. The three individual sessions are distributed at the beginning, middle, and towards the end of the training program. Individual Session 1 occurs after Group Session 1. It covers orientation to the training program, including orientation to and clarification of the Participant Handbook. Individual Session 2 occurs after Group Session 5 and involves review and implementation of training strategies. Individual Session 3 occurs after Group Session 9 and covers review of learned strategies, implementation of training strategies in daily life, and review of execution, obstacles, and adjustments required for individual projects.
  Arms: Cognitive Rehabilitation
Behavioral: Brain Health Education Program — The active control group will control for non-specific effects inherent to supervised CR. Participants will receive a manualized brain health education (BHE) training program, matched with the adapted CR intervention for therapist time and homework. Once these participants complete the 12 weeks of the control intervention and undergo the post-intervention assessments, participants will be offered the 12 weeks active intervention to ensure that all study participants have the potential of benefitting from CR.
  Arms: Brain Health Education Program

SUMMARY:
This pilot randomized controlled trial is to investigate the feasibility and efficacy of cognitive rehabilitation for patients with post-COVID-19 cognitive impairment. Additionally, the study will obtain preliminary data, using rsfMRI, regarding the potential underlying connectivity networks, mediating the effect of CR on cognitive improvements.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Have a confirmed SARS-CoV-2 infection (positive PCR or are serum antibody positive [against spike protein if unvaccinated or N-capsid peptide if vaccinated])
* Speak English
* Have objective mild to moderate cognitive impairment, which will be defined as impairment in executive function (a z-score >1.5 standard deviations below the normative mean) and in at least one other cognitive domain
* Endorse comfort and familiarity with technology.

Exclusion Criteria:

* No method of contact
* Major neurocognitive disorder, as defined by a score <17 on the Montreal Cognitive Assessment (MoCA)
* History of pre-COVID-19 neurologic disease (e.g., stroke)
* History of severe head injury (as defined by loss of consciousness >30 minutes)
* Ongoing substance use disorder (Mini International Neuropsychiatric Interview Version 7.0.2 [MINI] or Alcohol Use Disorders Test-Consumption [AUDIT-C] >8)
* Unstable medical, neurologic, or psychiatric conditions precluding participation in research activities, and
* Contraindication for MRI (e.g., metallic/electronic implants).
* Not involved in cognitive rehabilitation/training or daily meditative practices during study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Trail Making Test - Part B | end of study, at 12 months
  Trail Making Test - Part B: a measure of aspects of executive functioning (e.g., set- shifting and cognitive flexibility), where participants connect the dots on a page scattered with numbers and letters in alternating sequence. Scored by time in seconds. Higher number of seconds implies deficiencies in cognitive functioning.
Wisconsin Card Sorting Task (WCST)-64 | end of study, at 12 months
  Wisconsin Card Sorting Task (WCST)-64: Computer Version 2. The WCST-64 is a measure of executive functioning assessing novel problem solving and abstract thinking. The software scores the test and generates percentile scores (0-100). Scored by percentile. Higher percentile implies scoring better than others who have completed the task.
Acceptability Scale | end of study, at 12 months
  Acceptability: using 7 Likert-rated items (scores will be coded as: Low: ≤3; Moderate: 3-3.9; Good: ≥4).
  Full range from 1-7, with higher score indicating higher acceptability.
Enrollment yield | end of study, at 12 months
  Practicality measured by enrollment yield which is #enrolled/approached.
Dropout number | end of study, at 12 months
  Practicality measured by number of dropout
Staff Practicality | end of study, at 12 months
  Open-ended questions to staff regarding challenges conducting intervention (e.g., difficulty enrolling, reaching, engaging participants; scores will be coded as: Low: <50%; Moderate: 50-70%; Good: >70%).
Treatment Credibility and Expectancy Questionnaire. | end of study, at 12 months
  Participants' beliefs about how likely they are to benefit from the intervention using the Treatment Credibility and Expectancy Questionnaire. Full scale from 0-10, with higher score indicating higher treatment expectancy.
Resting state functional connectivity (rsFC) | end of study, at 12 months
  Neuroimaging Outcomes: Resting state functional connectivity (rsFC) within the central executive network (CEN).

SECONDARY OUTCOMES:
National Alzheimer's Coordinating Center (NACC) battery's Number Span | end of study, at 12 months
  Participants hear digit sequences of increasing lengths and have to recall them forward and in reversed order. Each level contains two equal number series with different numbers. Max score is 14 points for forward span and 14 points for backwards span. Higher score indicates better performance.
Paced Auditory Serial Addition Task (PASAT) | end of study, at 12 months
  Single digits are presented every 3 seconds and the participant must add each new digit to the one immediately prior to it. The score is the total number correct out of 60 possible answers. Full scale range from 0-60. Higher scores represent better performance.
Trail Making Test, Part A | end of study, at 12 months
  Requires participants to connect numbered dots in order as quickly as possible. A higher number of seconds implies worse performance.
The Symbol Digit Modalities Text (SDMT) | end of study, at 12 months
  Requires an individual to substitute digits for abstract symbols using a reference key as quickly as possible. Reaction times in seconds for the performance of the symbol-digit modalities test. A higher number of seconds implies worse performance.
The Hopkins Verbal Learning Test-Revised (HVLT-R) | end of study, at 12 months
  A list learning task that assesses learning (immediate recall) and memory (delayed recall) and recognition discrimination. The total score (higher score means a better outcome) is converted to a standardized "T" score using normative data. The possible "T" score for each participant ranges from 20 to 80, with higher scores indicative of better performance.
NACC battery's verbal phonemic and category fluency tests | end of study, at 12 months
  Requires participants to name as many words as they can beginning with a particular letter in 60 seconds, and then as many animals as they can, respectively. A higher number of words or animals named is indicative of better performance.
NACC battery's abbreviated Multilingual Naming Test (MINT) | end of study, at 12 months
  The MINT is a research measure intended to assess word retrieval deficits. It requires participants to name a series of individually presented line drawings that range from highly common (e.g. butterfly) to more obscure (e.g., axle) objects. The total scores range from 0 to 32, with higher scores indicating better performance.
Wide Range Achievement Test, reading subtest, 4th edition (WRAT-4) | end of study, at 12 months
  A measure of premorbid intellectual estimate. Scores range from 0-70, where a higher score indicates greater premorbid intellectual ability.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Wisnivesky, MD, DrPh, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. Any purpose. Data are available indefinitely at (Link to be included in the URL field below).

REFERENCES:
- [Derived] Becker JH, Watson E, Zubair N, Carnavali F, Bagiella E, Reich D, Wisnivesky JP. Preliminary evaluation of a cognitive rehabilitation intervention for post-COVID-19 cognitive impairment: A pilot randomized controlled trial. Neuropsychol Rehabil. 2025 Sep 24:1-12. doi: 10.1080/09602011.2025.2552154. Online ahead of print. PMID 40991647